CLINICAL TRIAL: NCT03392350
Title: Randomized Trial of the Impact of Body Scanning and Intensive Behavioral Intervention on Behavioral Change and Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reengineering Healthcare Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20111268
Record Dates: First submitted 2017-12-29; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Coronary Disease; Behavior and Behavior Mechanisms; Hypertension; Hypercholesterolemia
MeSH Terms: conditions — Coronary Disease; Behavior; Hypertension; Hypercholesterolemia | interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: One Control group one Intervention arm. The intervention group are the only subjects receiving a body scan consultation and behavioral intervention.
Who Masked: Investigator
Masking Description: The staff doing the end point assessment were blinded as to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Intervention arm (Active Comparator): A behavioral intervention consisting of a physician body scan consultation with a radiologist which included viewing self imagery followed by an 18 month behavioral intervention which included educational modules covering:
  Responding to Stress More Effectively Enhancing the effects of Relaxation Nourishing your immune system Energizing your Body Welcoming Others and Strengthening Relationships
  Interventions: Behavioral: Physician Body Scan Consultation with Behavioral Intervention
- Control Group (Active Comparator): No Intervention
  Interventions: Behavioral: Physician Body Scan Consultation with Behavioral Intervention

INTERVENTIONS:
Behavioral: Physician Body Scan Consultation with Behavioral Intervention — The RENEW™ program consisted of 7 bi-monthly face-to-face web sessions over 16-18 weeks followed by an average of 15 monthly check-in sessions (maintenance) over 80 weeks.This included modules on responding to stress, enhancing effects of relaxation, nourishing theimmune system, physical activity, and social support.

SUMMARY:
We evaluated the effectiveness of a combination of a comprehensive health assessment consisting of the combination of a screening full body scan employing graphic patient education and motivational techniques followed by intensive, individualized behavioral training and management program on improved adherence to beneficial lifestyle behaviors, as well as possibly reduced risk of disease.

DETAILED DESCRIPTION:
We initially enrolled 267 volunteer asymptomatic adults consisting of firefighters/police workers (n= 173), active military personnel (n= 57) and community college staff (n= 37). Subjects were randomized either to an intervention group or to usual care. The intervention group received The RENEW™ Program (www.therenewprogram.net) of lifestyle intervention as described below. A whole body CT scan was performed using a multidetector CT scan on all participants at baseline with the results discussed by a physician only in the intervention group, and after 2 years of follow-up a repeat scan was performed with a detailed evaluation of the results discussed by a physician with all participants (in part as a motivation to complete thestudy). This study was carried out in accordance with the recommendations of the Western Institutional Review Board with written informed consent from all subjects. All subjects gavewritten informed consent in accordance with the Declaration of Helsinki. The protocol wasapproved by the Western Institutional Review Board.

ELIGIBILITY:
Inclusion Criteria:

Men or women aged 35 and over who provide informed consent to participate including the baseline, interim, and follow-up clinic visits, as well as willingness to participate in the on-line intervention (if selected to be in that group) -

Exclusion Criteria:

Known cardiovascular disease, cancer, or any life-threatening or debilitating illness, including psychiatric illnesses, or significant difficulty with the English language that would preclude successful participation in the program

-

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2012-06-15 (Actual); Primary Completion 2015-09-15 (Actual); Study Completion 2015-11-20 (Actual)

PRIMARY OUTCOMES:
Progression of Coronary Artery Calcium | 2 years
  Coronary artery calcium (CAC) was assessed by a trained technologist with the Agatston score measured and volume score calculated, summed among the four major coronary arteries using conventional methods.

SECONDARY OUTCOMES:
Epicardial and Thoracic fat volume (in cm3) | 2 years
  The QFAT™ software was utilized to provide measures of epicardial and thoracic fat volume (in cm3) as described previously (20) in a subset of participants who had the required Dicom-archived CT scan data both pre and post intervention

IPD SHARING:
Plan to Share IPD: No